CLINICAL TRIAL: NCT01976039
Title: The Effectiveness of Rhinopharyngeal Retrograde Clearance on the Upper Airways Symptomatology and Function in Adults
Brief Title: Rhinopharyngeal Retrograde Clearance is Effective to Adequate Upper Airways Function in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Naomi Kondo Nakagawa, Associate Professor of Faculdade de Medicina da Universidade de São Paulo, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEP-FMUSP 211-11
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Nasal Obstruction; Exposure to Pollution
Keywords: motorcyclist; nasal mucociliary clearance; physical therapy
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RRC (Other): rhinopharyngeal retrograde clearance (RRC) isolated: First patient sits in a chair. Second: patient inhales air deeply and exhales making noise and vibration in the upper airway to facilitate swalling. Third patients finishes with another deep inhalation. This technique is new, simple to use and with no cost. No need of any material or equipment.
  Interventions: Other: rhinopharyngeal retrograde clearance (RRC)
- RRC+S (Experimental): retrograde rhinopharyngeal retrograde clearance combined with saline instillation (RRC+S): patient sits in a chair and inhaled air and make noise and vibrate the upper airway at the same instills saline into the nare to facilitate nose washing and swalling. This technique is new, simple to use and with low cost (only saline).
  Interventions: Other: rhinopharyngeal retrograde clearance (RRC)

INTERVENTIONS:
Other: rhinopharyngeal retrograde clearance (RRC) — The rhinopharyngeal retrograde clearance is a respiratory physical therapy technique that uses a forced inspiratory maneuver to clear the nasopharynx with the aid of saline instillation
  Other Names: RCC+S

SUMMARY:
Professionals working in polluted areas may present increased clinical airways symptoms and dysfunction. Rhinopharyngeal retrograde clearance (RRC) has been used to improve mucus clearance in infants with bronchitis and bronchiolitis, and instillation the nasal cavity with saline has been used to reduce nasal inflammation in rhinitis and sinusopathies. The aim of this study was to assess the effects of RRC and RCC combined with saline (RRC+S) on nasal mucociliary clearance (MCC), mucus surface property, cellularity and airways symptoms in professional motorcyclists.

DETAILED DESCRIPTION:
Male motorcyclists (mean age 36 years) were recruited and randomly assigned to RRC or RRC+S. Subjects were assessed at baseline and 15 days after interventions for saccharin test, mucus contact angle, cellularity in nasal lavage and airways symptoms with the use of SNOT-20 questionnaire. Data were analyzed by two-way ANOVA for repeated measures with Bonferroni´s correction. A passive monitoring-system of nitrogen dioxide was used to assess the individual air pollution exposure along the study period. The association between nitrogen dioxide and the airways outcomes was analyzed by Spearman correlation test.

ELIGIBILITY:
Inclusion Criteria:

* Professional motorcyclists aged 18 years to 45 years
* Minimum of one year in that occupation
* Agreement with the written informed consent

Exclusion Criteria:

* Smokers
* Inability to understand and to follow commands
* Previous nasal surgery
* Respiratory infection in the previous 30 days

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Saccharine transit time test (STT) | 15 days
  To measure nasal mucociliary clearance. Subjects were asked to report the first perception of a sweet taste after 25 mg of saccharine powder was deposited in the free airflow nostril.

SECONDARY OUTCOMES:
mucus surface property | 15 days
  The contact angle of nasal mucus was measured.

OTHER OUTCOMES:
SNOT-20 | 15 days
  A questionnaire to assess the symptoms of the nose and airways for rhinosinusitis

CONTACTS AND LOCATIONS:
Overall Officials: Naomi K Nakagawa, PhD, Principal Investigator — University of Sao Paulo; Paulo HN Saldiva, PhD, Study Director — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Faculdade de Medicina da Universidade de São Paulo, São Paulo

REFERENCES:
- [Background] Gomes EL, Postiaux G, Medeiros DR, Monteiro KK, Sampaio LM, Costa D. Chest physical therapy is effective in reducing the clinical score in bronchiolitis: randomized controlled trial. Rev Bras Fisioter. 2012 Jun;16(3):241-7. doi: 10.1590/s1413-35552012005000018. Epub 2012 Apr 12. PMID 22499404
- [Background] Proenca de Oliveira-Maul J, Barbosa de Carvalho H, Goto DM, Maia RM, Flo C, Barnabe V, Franco DR, Benabou S, Perracini MR, Jacob-Filho W, Saldiva PHN, Lorenzi-Filho G, Rubin BK, Nakagawa NK. Aging, diabetes, and hypertension are associated with decreased nasal mucociliary clearance. Chest. 2013 Apr;143(4):1091-1097. doi: 10.1378/chest.12-1183. PMID 23100111
- [Background] Piccirillo JF, Merritt MG Jr, Richards ML. Psychometric and clinimetric validity of the 20-Item Sino-Nasal Outcome Test (SNOT-20). Otolaryngol Head Neck Surg. 2002 Jan;126(1):41-7. doi: 10.1067/mhn.2002.121022. PMID 11821764
- [Background] Belda J, Parameswaran K, Keith PK, Hargreave FE. Repeatability and validity of cell and fluid-phase measurements in nasal fluid: a comparison of two methods of nasal lavage. Clin Exp Allergy. 2001 Jul;31(7):1111-5. doi: 10.1046/j.1365-2222.2001.01133.x. PMID 11468003
- [Background] Nakagawa NK, Franchini ML, Driusso P, de Oliveira LR, Saldiva PH, Lorenzi-Filho G. Mucociliary clearance is impaired in acutely ill patients. Chest. 2005 Oct;128(4):2772-7. doi: 10.1378/chest.128.4.2772. PMID 16236954
- [Background] Cancado JE, Braga A, Pereira LA, Arbex MA, Saldiva PH, Santos Ude P. [Clinical repercussions of exposure to atmospheric pollution]. J Bras Pneumol. 2006;32 Suppl 2:S5-11. doi: 10.1590/s1806-37132006000800003. Portuguese. PMID 17273599
- [Derived] Brant TC, Yoshida CT, Carvalho Tde S, Nicola ML, Martins JA, Braga LM, Oliveira RC, Leyton V, Andre CS, Saldiva PH, Rubin BK, Nakagawa NK. Mucociliary clearance, airway inflammation and nasal symptoms in urban motorcyclists. Clinics (Sao Paulo). 2014;69(12):867-70. doi: 10.6061/clinics/2014(12)13. PMID 25628001